CLINICAL TRIAL: NCT05585515
Title: Study of Identification of Metabolomics-based Sleepiness Markers for Risk Prevention and Traffic Safety
Brief Title: Metabolomics-based Sleepiness Markers
Acronym: ME-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Fonds für Verkehrssicherheit FVS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-01273; SNCTP000005089 (Registry Identifier: Swiss National Clinical Trials Portal)
Record Dates: First submitted 2022-10-05; First posted 2022-10-18 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Sleep Deprivation; Sleepiness; Insufficient Sleep Syndrome
Keywords: metabolomics; sleep; biomarker; impairment
MeSH Terms: conditions — Sleep Deprivation; Sleepiness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): 16/8 hours wake/sleep regime for 3 consecutive days at home and for consecutive 2 days in sleep laboratory
- Sleep restriction (Experimental): 18/6 hours wake/sleep regime for 3 consecutive days at home and one day in sleep laboratory, followed by recovery night of 8 hours sleep
  Interventions: Behavioral: Sleep restriction
- Sleep deprivation (Experimental): 16/8 hours wake/sleep regime for 3 consecutive days at home, one night of sleep deprivation (24/0 hours) in sleep laboratory, followed by recovery night of 8 hours sleep
  Interventions: Behavioral: Sleep deprivation

INTERVENTIONS:
Behavioral: Sleep deprivation — Total sleep deficit of consecutive 8 hours
  Arms: Sleep deprivation
Behavioral: Sleep restriction — Total sleep deficit of cumulative 8 hours
  Arms: Sleep restriction

SUMMARY:
Estimating that people sleep on average up to two hours less over the last decades, sleepiness and fatigue need to be considered as significant societal problems of the modern world. Jurisdiction is precise on how to deal with overtired offenders since they were not allowed to use machines or vehicles in the first place, similar to drunk individuals or consumers of illicit drugs. In contrast to alcohol or illicit drug use, however, there are no quick roadside or workplace tests as objective (analytical) biomarkers for sleepiness.

Investigators hypothesize that increasing sleep drive or impaired wakefulness can be assessed by qualitative or quantitative fluctuations of certain metabolites in biological specimens, e.g., accumulation or decrease of endogenous substances related to sleep debt. Thus, this sleep study provides the necessary biological samples of either sleep-deprived, sleep-restricted, or control subjects, which are then analysed for appropriate metabolite biomarkers utilizing an untargeted metabolomics approach. In addition to established impairment tests, a state of the art driving simulator will be employed to objectively measure driving performance under all study conditions. Participants will also rate their subjective sleepiness using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* understanding and spoken command of German language
* good health condition
* Body Mass Index between 18.5-24.9 kg/m2
* habitual average sleep duration between 7-9 hours / night
* habitual consumption of 3 or fewer caffeinated beverages / day
* habitual consumption of 5 or fewer alcoholic beverages / week
* good sleep quality: Pittsburgh Sleep Quality Index score ≤ 5
* reasonable oral hygiene (≥1 tooth brushing / day)
* normal or corrected-to-normal vision
* car driving license holder since at least 2 years (obtained in a country with right hand traffic) and regular driver (≥ 1 per week)

Exclusion Criteria:

* two or more time zone crossings in the last 3 months
* habitual napper
* history or presence of neurological disorder, psychiatric disorder, cardiovascular disorder, dental disorder or any disorder that could pose a risk in participating or that could possibly influence study measurements
* history or presence of a sleep disorder (screening night)
* use of illicit drugs (urinary drug screening)
* use of current medication (urinary drug screening) known to influence study measurements
* extreme chronotype (reduced Morningness-Eveningness-Questionnaire score ≤7 or ≥22)
* current smoker
* habitual use of energy drinks (>1 / week)
* severe skin allergies or hypersensitivities
* food allergies
* hospital stay in past 6 months
* shift worker, night worker
* recent past (last 3 months) or present Covid-19 infection
* fainting at the sight of blood or needles
* participation in a clinical study less than 30 days ago or is currently participating in other clinical studies
* simulator sickness syndrome
* refusal to sign informed consent

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Changes in metabolite concentrations in oral fluid quantified by liquid chromatography with mass spectrometry | After arrival at study site (6pm, baseline), repeatedly during scheduled wakefulness (8am, 12pm, 4pm, 7pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  Investigators will collect oral fluid samples from participants for quantification of all detectable metabolites. Investigators will analyze which metabolite concentration values undergo significant changes during sleep deficit conditions in comparison to control condition and also show effects of recovery sleep. These will serve as candidate biomarkers.

SECONDARY OUTCOMES:
Driving performance | morning after experimental night (10am)
  Investigators will gather driving simulation results via Standardized Application for Fitness to Drive Evaluations (S.A.F.E. scale), and analyze their changes after sleep deficit in comparison to control condition. This scale has a range from 0 (best) to 10 (worst) in full steps.
Psychomotor Vigilance Test | After arrival at study site (6pm, baseline), repeatedly during scheduled wakefulness (8am, 12pm, 4pm, 7pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  The Psychomotor Vigilance Test is a gold standard reaction time test to assess vigilance and sustained attention.
d2 Test of Attention | After arrival at study site (6pm, baseline), repeatedly during scheduled wakefulness (8am, 12pm, 4pm, 7pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  The d2 Test of Attention is a paper and pencil test to assess selective and sustained attention and visual scanning speed.
Visual attention test | After arrival at study site (8pm, baseline), repeatedly during scheduled wakefulness (10am, 2pm, 6pm, 8pm), and morning after recovery night of 8 hours of sleep (8am)
  The visual attention test is a virtual reality glasses test to assess visual skills in a complex visual environment.
Subjective situational sleepiness | After arrival at study site (6pm, baseline), repeatedly during scheduled wakefulness (8am, 12pm, 4pm, 7pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  Participants will complete the Karolinska Sleepiness Scale questionnaire.
Subjective sleepiness | After arrival at study site (6pm, baseline), repeatedly during scheduled wakefulness (8am, 12pm, 4pm, 7pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  Participants will complete the Stanford Sleepiness Scale questionnaire.
Electroencephalographic changes | During scheduled sleep, driving simulation test (10am), and at two time points during scheduled wakefulness (12pm, 7pm)
  Investigators will analyze changes in sleep and wake electroencephalographic patterns of participants by calculating sleep scores according to American Academy of Sleep Medicine (AASM) scoring manual.
Behavioral markers of drowsy driving | Once per study arm after driving simulation test (11am)
  Investigators will examine participants after driving simulation test for behavioral abnormalities concerning orientation, coordination, speech, mood, appearance, reaction, and pupillary light reflex.
Changes in metabolite concentrations in exhaled breath quantified by liquid chromatography with mass spectrometry | After arrival at study site (8pm, baseline), repeatedly during scheduled wakefulness (10am, 2pm, 6pm, 8pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  Investigators will collect exhaled breath samples from participants for quantification of all detectable metabolites. Investigators will analyze which metabolite concentration values undergo significant changes during sleep deficit conditions in comparison to control condition and also show effects of recovery sleep. These will serve as secondary candidate biomarkers.
Changes in metabolite concentrations in finger sweat quantified by liquid chromatography with mass spectrometry | After arrival at study site (8pm, baseline), repeatedly during scheduled wakefulness (10am, 2pm, 6pm, 8pm, 11pm), and morning after recovery night of 8 hours of sleep (8am)
  Investigators will collect finger sweat samples from participants for quantification of all detectable metabolites. Investigators will analyze which metabolite concentration values undergo significant changes during sleep deficit conditions in comparison to control condition and also show effects of recovery sleep. These will serve as secondary candidate biomarkers.
Correlation of metabolic changes between blood and non-invasive specimens | immediately after driving simulation test (11am)
  Investigators will compare metabolite concentrations in non-invasive matrices (oral fluid, finger sweat, exhaled breath, and dried blood spots) and compare those with blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Keller, Dr, Principal Investigator — University of Zurich, Zurich
Locations (1):
- Human Sleep Laboratory, University of Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in peer-reviewed journals. Anonymized raw data will be made available upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: starting after publication
Access Criteria: upon request via e-mail

REFERENCES:
- [Derived] Scholz M, Lakaemper S, Keller K, Dobay A, Steuer AE, Landolt HP, Kraemer T. Metabolomics-based Sleepiness Markers for Risk Prevention and Traffic Safety (ME-SMART): a monocentric, controlled, randomized, crossover trial. Trials. 2023 Feb 21;24(1):131. doi: 10.1186/s13063-023-07154-x. PMID 36810100